CLINICAL TRIAL: NCT05597670
Title: Effect of Proximal Stabilization on Recruitment of the Core & Vasti in Patients With Patellofemoral Arthritis as They Descend Stairs
Brief Title: Effect of Proximal Stabilization on Recruitment of the Core & Vasti in Patellofemoral Arthritis During Descending Stairs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Jilan Adel yousef, lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P.T.REC/012/003438
Record Dates: First submitted 2022-10-25; First posted 2022-10-28 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Chondromalacia Patellae
MeSH Terms: conditions — Chondromalacia Patellae

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned into two groups, group A and group B . Patients in both groups will receive a traditional physical therapy treatment, but group (B) will receive additional proximal stability exercise.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Other): Patients in this group will receive a traditional therapeutic knee rehabilitation program in the form of mini-squatting exercise (up to 45 degree knee flexion measured by a universal goniometer) , strengthening of hip abductors and external rotators
  Interventions: Other: traditional knee rehabilitation program
- group B (Experimental): Patients in this group will receive the same program as group (A) plus proximal stabilization exercise
  Interventions: Other: traditional knee rehabilitation program; Other: proximal stabilization

INTERVENTIONS:
Other: traditional knee rehabilitation program — Patients in this group will receive a traditional therapeutic knee rehabilitation program in the form of mini-squatting exercise (up to 45 degree knee flexion measured by a universal goniometer) , strengthening of hip abductors and external rotators
Other: proximal stabilization — the principles of proximal stability will be explained to patients before initiation of treatment and patients will be asked to comply with these principles during exercise. These principles include learning how to activate transversus abdominus by abdominal bracing without allowing pelvis tilting and ensure neutral spine and diaphragmatic breathing during exercise.
  Arms: group B

SUMMARY:
Purpose: to investigate the effect of proximal stability on PF OA. Methods: Thirty patients with PF OA will be recruited. Patients will be randomly assigned into two groups, group A and group B . Patients in both groups will receive a traditional physical therapy treatment, but group (B) will receive additional proximal stability exercise. All patients will be evaluated for muscular recruitment strategies (onset and duration) of multifidus, transversus abdominus (TrA), gluteus medius (GM), and vasti measured by quantitative Electromyography during stair descent. pre and post-treatment.

DETAILED DESCRIPTION:
: A) Procedures for evaluation: The practical section of the studywill be undertaken in 6 weeks (2 sessions a week). Measurement will be taken before the start of treatment program then after the end of 6 weeks treatment program. Investigators will collect the EMG activity of VMO, VL, GM, multifidus, and TrA using bipolar Ag-AgCl disposable surface electrodes (Better signal solution medical supply Co., limited, Zhongshan, China) and eight channels highresolution wireless bio amplifier (WBA) system (Biomation, Almonte, Canada). Electromyographic data will be sampled at 1000 Hz and bandpass filtered at 50-200 Hz. For each muscle, three electrodes will be used; two electrodes will be placed ~ 30 mm apart in the direction of the muscle fibers and a ground electrode will be placed over the closest bony prominence. Before placement of the electrodes, the subject's skin will be cleaned with alcohol to reduce impedance and excess hair will be removed to eliminate shifting of the electrodes if needed. The stairstepping task will consist of descending 2 steps Before data acquisition, participants will be asked to perform one practice trial of stair descent to get familiarized with the task. Then the participants will perform three test trials with thirty seconds of rest after each trial to prevent fatigue. The raw data will be stored on a personal computer for analysis with a custom program in Matlab . Investigators will use a mean of data in three trials for analysis.

b) Procedures for treatment: All patients will receive a traditional physical therapy program in the form of TENS , stretching hamstring, quadriceps and calf muscles

* Group (A) Patients in this group will receive a traditional therapeutic knee rehabilitation program in the form of mini-squatting exercise (up to 45 degrees knee flexion measured by a universal goniometer) , strengthening of hip abductors and external rotators using clamshell exercise . No emphasis will be placed on stabilizing the core musculature before initiating any of those exercises.
* Group (B) Patients in this group will receive the same program as group (A) plus proximal stability exercise and the principles of proximal stability will be explained to patients before initiation of treatment and patients will be asked to comply with these principles during exercise. These principles include learning how to activate transversus abdominus by abdominal bracing without allowing pelvis tilting and ensure neutral spine and diaphragmatic breathing during exercise.

ELIGIBILITY:
Inclusion Criteria:

1. Anterior- or retro-patellar knee pain aggravated by at least two activities that load the PFJ (eg; stair ambulation, squatting and/or rising from sitting) .
2. Pain during these activities presented on most days during the past month and their pain severity was ≥ 4 on an 11 point numerical pain scale during aggravating activities .,
3. A grade less than (2) from postero-anterior views on the Kellgren - Lawrence (KL) grading scale.

Exclusion Criteria:

1. concomitant pain from tibiofemoral joint or other knee structures .
2. current or previous pain in the hip, lumbar spine or foot that had lasted longer than 3 months and/or required intervention.
3. a history of lower extremity, pelvis or spine fractures; spine, hip, knee or foot surgeries; hip or patellar subluxation/ dislocation.
4. injury to any of knee ligaments or meniscus.
5. systemic diseases (e.g. rheumatoid arthritis), neurological conditions or fibromyalgia .
6. The professional athletes; people who exercise more than two hours a day or every other day, will be excluded.

Ages: 35 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-11-29 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
The change of EMG onset of multifidus | baseline and six weeks
  investigators will collect the EMG activity of multifidus by electromyography (EMG) using surface electrodes
The change of EMG duration of multifidus | baseline and six weeks
  investigators will collect the EMG activity of multifidus by electromyography (EMG) using surface electrodes
The change of EMG duration of vastus medialis obliqus | baseline and six weeks
  investigators will collect the EMG activity of vastus medialis obliqus by electromyography (EMG) using surface electrodes
The change of EMG onset of vastus medialis obliqus | baseline and six weeks
  investigators will collect the EMG activity of vastus medialis obliqus by electromyography (EMG) using surface electrodes
The change of EMG onset of vastus lateralis | baseline and six weeks
  investigators will collect the EMG activity of vastus lateralis by electromyography (EMG) using surface electrodes
The change of EMG duration of vastus lateralis | baseline and six weeks
  investigators will collect the EMG activity of vastus lateralis by electromyography (EMG) using surface electrodes
The change of EMG duration of gluteus medius | baseline and six weeks
  investigators will collect the EMG activity of gluteus medius by electromyography (EMG) using surface electrodes
The change of EMG onset of gluteus medius | baseline and six weeks
  investigators will collect the EMG activity of gluteus medius by electromyography (EMG) using surface electrodes
The change of EMG onset of transversus abdominus | baseline and six weeks
  investigators will collect the EMG activity of transversus abdominus by electromyography (EMG) using surface electrodes
The change of EMG duration of transversus abdominus | baseline and six weeks
  investigators will collect the EMG activity of transversus abdominus by electromyography (EMG) using surface electrodes

SECONDARY OUTCOMES:
kinesiophobia | baseline and six weeks
  patients will respond to the questions of the Tempa scale

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of physical therapy, Cairo university, Giza, Egypt